CLINICAL TRIAL: NCT03011671
Title: A Phase I Study of Safety and Tolerability of Acetazolamide With Temozolomide in Adults With Newly Diagnosed MGMT Promoter-Methylated IDH Wildtype Glioblastoma
Brief Title: Study of Acetazolamide With Temozolomide in Adults With Newly Diagnosed or Recurrent Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB16-0767
Record Dates: First submitted 2017-01-04; First posted 2017-01-05 (Estimated); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Malignant Glioma of Brain
Keywords: Malignant Glioma of Brain; Acetazolamide; Temozolomide
MeSH Terms: interventions — Acetazolamide; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Acetazolamide with Temozolomide (Experimental): Subjects will receive daily ACZ together with TMZ in 28 day cycles for up to 6 cycles if they do not experience either disease worsening or unacceptable side effects.
  Interventions: Drug: Acetazolamide; Drug: Temozolomide

INTERVENTIONS:
Drug: Acetazolamide — ACZ will be given at an initial dose of 250 mg twice a day (BID) and then escalated to 500 mg BID after 1 week. ACZ will be given on days 1-21 of each cycle.
  Other Names: Diamox; Diamox Sequels
Drug: Temozolomide — For cycle 1 of the maintenance phase, TMZ will administered at 150 mg/m2 on days 1- 5 followed by 23 days with no drug. For cycles 2- 6, TMZ can be increased to 200 mg/m2 at the discretion of the treating investigator.
  Other Names: Temodar

SUMMARY:
This is a Phase I study that examines the rate of dose limiting side effects in patients with malignant astrocytoma treated with combination acetazolamide (ACZ) and temozolomide (TMZ). Eligible patients must have histologically proven newly diagnosed, O6-methylguanine-DNA methyltransferase (MGMT) methylated WHO grade III or IV astrocytoma and be planning to undergo treatment with standard adjuvant TMZ (after completing treatment with TMZ and ionizing radiation (IR)).

During this study, patients will receive daily oral ACZ with TMZ. During each cycle, ACZ will be started on the day of TMZ initiation and continued for a total of 21 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven, newly diagnosed IDH wildtype glioblastoma (GBM) that has a methylated MGMT promoter as assessed by the standardized institutional analysis.
* Patients are eligible if they had a prior low grade astrocytoma and there is subsequent histological evidence of a diagnosis of grade III or IV tumor.
* Patients must be receiving TMZ as part of their standard adjuvant treatment regimen following treatment with TMZ and Radiation.
* Patients must have a Karnofsky performance ≥ 60%.
* Normal organ function as follows:

  * Absolute Neutrophil Count (ANC) ≥ 1.0 x 10^9/ L
  * Platelets ≥ 100 x 10^9 / L
  * Hemoglobin ≥ 8.0 g / dL
* Age 18 years or older.
* Kidney function (creatinine level within normal institutional limit, or creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine level above institutional normal).
* Liver function (AST/ALT <2.5 X institutional upper limit of normal (ULN), Total bilirubin ≤ 1.5 times ULN, INR within 1.5 times ULN (or if receiving anticoagulant therapy an INR of ≤ 3.0 is allowed with concomitant increase in PT or an aPTT ≤ 2.5 × control).
* Women able to become pregnant must have a negative pregnancy test within 30 days of registration.
* Patients must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior invasive malignancy that is not low-grade glioma (except non-melanomatous skin cancer or carcinoma in situ of the cervix) unless the patient has been disease free and off therapy for that disease for a minimum of 3 years.
* Active systemic infection requiring treatment, including any HIV infection or toxoplasmosis.
* Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration.
* Systemic corticosteroid therapy, >8 mg of dexamethasone daily (or equivalent) at study enrollment.
* Pregnant women are excluded from this study, where pregnancy is confirmed by a positive serum beta-hCG laboratory test. Breast-feeding should be discontinued.
* Hypersensitivity to acetazolamide or sulfonamides.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 28 Days
  To determine the safety, tolerability and adverse event profile of adding acetazolamide to temozolomide in patients with newly diagnosed malignant astrocytoma.

SECONDARY OUTCOMES:
Measure objective response rate (ORR); change in tumor size | 6 months
  ORR will be determined at 6 months and is based on the change in tumor size (as determined by Response Assessment in Neuro-Oncology Criteria (RANO) criteria) at the indicated time relative to the pre-treatment scan. RANO criteria will also be used to define disease status (CR, PR, etc.).
Time until progression free survival (PFS) | 6 months
Time until overall survival (OS) | From start date of therapy to the date of death from any cause, whichever may come first, assessed up to 100 months
Analysis of formalin fixed paraffin embedded surgical specimens. | Through study completion an average of one year
  Bcl-3 expression will be determined by an independent neuro-pathologist by immunohistochemical analysis of formalin fixed paraffin embedded (FFPE) surgical specimens. This is to evaluate Bcl-3 expression level within each tumor and preliminarily examine the ability of Bcl-3 to predict response to TMZ and the efficacy of adding ACZ.
To determine feasibility of cooperative interaction between multiple sites | End of study enrollment period (approximately 6 years)
  Feasibility to be determined based on ability to complete accrual to the study

CONTACTS AND LOCATIONS:
Overall Officials: Bakhtiar Yamini, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States